CLINICAL TRIAL: NCT00185393
Title: Efficacy and Safety of Subsequent Treatment With [90]Y-Ibritumomab Tiuxetan Versus no Further Treatment in Patients With Stage III or IV Follicular Non-Hodgkin's Lymphoma Having Achieved Partial or Complete Remission After First Line Chemotherapy. A Prospective, Multicenter, Randomized Phase III Clinical Trial
Brief Title: Treatment With [90]Y-Ibritumomab Tiuxetan Versus no Treatment in Patients With Follicular Non Hodgkin Lymphoma (Stage III or IV) Having Achieved a Partial or Complete Remission After First Line Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90966; 304820; NHL FIT
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Follicular Non Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Biological: Zevalin ([90]Y-ibritumomab tiuxetan, BAY86-5128)
- Arm 2 (Other)
  Interventions: Other: no treatment

INTERVENTIONS:
Biological: Zevalin ([90]Y-ibritumomab tiuxetan, BAY86-5128) — treatment with 90 Yttrium-labeled anti CD 20 antibody
  Arms: Arm 1
Other: no treatment — no treatment
  Arms: Arm 2

SUMMARY:
The aim of the study is to test [90]Y-ibritumomab tiuxetan, a radioactive antibody, in patients with stage III or IV follicular lymphoma whose disease is in partial or complete remission after first line chemotherapy. The radioactive antibody will be compared with no further treatment to see which is better in the long term after standard lymphoma treatment.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Non Hodgkin Lymphoma stage III or IV at timepoint of diagnosis
* Patients who have achieved a remission after first line chemotherapy
* No less than 6 weeks and no more than 12 weeks since last dose of chemotherapy
* older than 18 years
* written informed consent

Exclusion Criteria:

* Any other anticancer treatment for NHL except the preceding first line chemotherapy
* Prior radiation therapy
* Patients who have not recovered from the toxic effects of the first line chemotherapy
* Any other cancer or history of cancer less than 10 years ago
* Patients with known HIV positivity
* patients with pleural effusion or ascites
* female patients who are pregnant or breast feeding (women of childbearing potential must have a negative serum pregnancy test at study entry)
* Adults not employing an effective method of birth control during study treatment and 12 months thereafter
* Patients unable or unwilling to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2001-08; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Progression free survival | End of study

SECONDARY OUTCOMES:
Clinical and molecular response rates | End of study
Overall survival | End of study
Quality of Life | End of study
Adverse events / Toxicity Grading | Continous
Clinical laboratory results | 3 monthly
Vital signs / physical examination | 3 monthly
ECG | End of study
Co-medication | Continous

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (87):
- Belgium (6):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Leuven
  - Yvoir
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Denmark (2):
  - Aarhus
  - Copenhagen
- France (14):
  - Rennes, Brittany Region
  - Angers
  - Besançon
  - Bordeaux
  - Créteil
  - Grenoble
  - Le Mans
  - Lille
  - Lyon
  - Paris
  - Pierre-Bénite
  - Rouen
  - Strasbourg
  - Tours
- Germany (10):
  - Tübingen, Baden-Wurttemberg
  - Augsburg, Bavaria
  - München, Bavaria
  - Göttingen, Lower Saxony
  - Münster, Nordrhein-Westfalen / 298
  - Hamm, Nordrhein-Westfalen / 358
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Dresden, Saxony
  - Hamburg
- Italy (10):
  - Bologna, BO
  - San Giovanni Rotondo, Foggia
  - Milan, MI
  - Rozzano, MI
  - Pisa, PI
  - Roma, Roma
  - Torino, TO
  - Milan
  - Napoli
  - Palermo
- Netherlands (12):
  - Amersfoort
  - Amsterdam
  - Eindhoven
  - Enschede
  - Groningen
  - Leiden
  - Maastricht
  - Nijmegen
  - Rotterdam
  - The Hague
  - Utrecht
  - Zwolle
- Norway (2):
  - Oslo
  - Tromsø
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Spain (6):
  - L'Hospitalet de Llobregat, Barcelona
  - Barcelona
  - Madrid
  - Málaga
  - Salamanca
  - Valencia
- Sweden (3):
  - Gothenburg
  - Umeå
  - Uppsala
- Switzerland (7):
  - Zurich, Bern / 633
  - Sankt Gallen, Saint Gallen / 633
  - Aarau
  - Bellinzona
  - Bern
  - Geneva
  - Lausanne
- United Kingdom (6):
  - Glasgow
  - London
  - Manchester
  - Newcastle upon Tyne
  - Plymouth
  - Surrey